CLINICAL TRIAL: NCT04067102
Title: Albumin Bound (Nab)-Paclitaxel Combined With Carboplatin Versus Paclitaxel Combined With Carboplatin Followed by Epirubicin and Cyclophosphamide as Neoadjuvant Treatment for Participants With Triple Negative Breast Cancer (TNBC)
Brief Title: Nab-paclitaxel Based Regimens VS Paclitaxel Based Regimens in Neoadjuvant Treatment for TNBC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruited
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Liu Yunjiang, Professor, Director and Vice-president, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNBC-NEO
Record Dates: First submitted 2019-08-14; First posted 2019-08-26 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-paclitaxel Based Regimens (Experimental)
  Interventions: Drug: Albumin bound (nab)-paclitaxel combined with carboplatin followed by epirubicin and cyclophosphamide
- Paclitaxel Based Regimens (Active Comparator)
  Interventions: Drug: paclitaxel combined with carboplatin followed by epirubicin and cyclophosphamide

INTERVENTIONS:
Drug: Albumin bound (nab)-paclitaxel combined with carboplatin followed by epirubicin and cyclophosphamide — Paclitaxel for injection (albumin binding)260mg/m2，I.v., d1；carboplatin AUC=5, I.v., d1； 21 days in one cycle, 4 cycles in total.Continue the protocol when evaluated as CR/PR/SD at the second cycle, Terminate the protocol paclitaxel (albumin binding) combined with carboplatin when evaluated as PD at the second cycle，and use the EC protocol in advance or decide the next treatment
  Arms: Nab-paclitaxel Based Regimens
Drug: paclitaxel combined with carboplatin followed by epirubicin and cyclophosphamide — Paclitaxel 175mg/m2, I.v., d1； Carboplatin injection AUC 5, I.v., d1； 21 days in one cycle, 4 cycles in total.Continue the protocol when evaluated as CR/PR/SD at the second cycle, Terminate the protocol paclitaxel (albumin binding) combined with carboplatin when evaluated as PD at the second cycle，and use the EC protocol in advance or decide the next treatment protocol by the researcher
  Arms: Paclitaxel Based Regimens

SUMMARY:
To evaluate the efficacy and safety of P nab-paclitaxel combined with carboplatin versus paclitaxel combined with carboplatin followed by epirubicin and cyclophosphamide in the neoadjuvant treatment of triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥ 18 yrs and ≤70 yrs；
* Histological confirmation of Unilateral primary invasive breast cancer, cT2-4NanyM0, planning to receive neoadjuvant chemotherapy；
* The expression of ER<10%，PR <10% and Her-2 negative by immunohistochemical, if HER2 expression ++, further FISH test confirmed no amplification of Her-2 gene；
* ECOG performance status 0-1；
* LVEF≥55%；
* Bone marrow function: neutrophils ≥ 1.5×109/L, platelets ≥ 100×109/L, hemoglobin ≥ 90 g/L；
* Liver and renal function：Serum creatinine ≤ 1.5x ULN；Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN；Total bilirubin ≤ 1.5x ULN or when patients with Gilbert's syndrome ≤ 2.5x ULN；
* The patient has good compliance with the planned treatment, understands the research process of the study and signs a written informed consent form.

Exclusion Criteria:

* Cytotoxic chemotherapy, endocrine therapy or radiation therapy for any reason；
* New York Heart Association (NYHA) score identifies patients with heart disease above grade II (including grade II)；
* Patients with severe systemic infections or other serious illnesses；
* Patients known to be allergic or intolerant to chemotherapeutic drugs or their excipients；
* Combined with other malignant tumors or had malignant tumors other than breast cancer in the past 5 years, except for cervical carcinoma in situ and non-melanoma skin cancer that have been fully treated；
* Women of childbearing age who are pregnant or lactating and who refuse to take appropriate contraceptive measures during the trial；
* Participated in other experimental studies within 30 days before the first dose of study drug administration
* Researchers judged patients who were unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（pCR） | 6 months
  pCR is defined as no histologic evidence of invasive tumor cells in the surgical breast specimen, axillary nodes, or sentinel node identified after neoadjuvant chemotherapy (ypT0/Tis ypN0)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 months
  Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR)
Disease-free survival（DFS） | 5 years
  Disease-free survival refers to the time from surgical resection of breast cancer to clinically confirmed local recurrence, distant metastasis, second primary tumor diagnosis, or patient death.
Overall survival（OS） | 5 years
  Overall survival is defined as the length of time from random assignment to death or to last contact.
adverse events（AEs） | until 28 days after the last study drug administration
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Yunjiang Liu, MD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China